CLINICAL TRIAL: NCT00506480
Title: Phase 1 Study of Endometrial Markers of Endometrial Receptivity in Oocyte Donation
Brief Title: Assessment of Endometrial Receptivity in Recipients of Donated Oocytes
Acronym: ERPOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 319-08.07
Record Dates: First submitted 2007-07-22; First posted 2007-07-25 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2007-07

CONDITIONS: Embryo Implantation
Keywords: Embryo Implantation; Endometrium; endometrial implantation; Oocyte Donation; in vitro fertilization; endometrial sampling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OD (Experimental): patients artificially prepared for OD will undergo a mock cycle consisting of estrogen and later by progesterone. a pipelle sample will be taken after 6 days of progesterone supplementation.
  Interventions: Procedure: endometrial sampling
- IVF (Experimental): A pipelle sample will be taken on day 21 of the cycle before administration of GNRHa. Exact timing will be performed by counting 7 days from the LH surge.
  Interventions: Procedure: endometrial sampling

INTERVENTIONS:
Procedure: endometrial sampling — Endometrial biopsy is a procedure in which a tissue sample is obtained from the endometrium. This procedure is performed without anesthesia during pelvic examination. The cervix is cleaned with an antiseptic solution and then grasped with an instrument (tenaculum) to steady the uterus. A small, hollow plastic tube is gently passed into the uterine cavity. Gentle suction removes a sample of the lining. The tissue sample and instruments are removed, and the sample is examined by pathology, immunohistochemistry, PCR and western blotting.

SUMMARY:
The purpose of this study is to determine whether endometrial receptivity markers obtained by endometrial sampling are effective in prediction of in vivo human embryo implantation.

DETAILED DESCRIPTION:
Since the introduction of In vitro fertilization (IVF), substantial improvements have been developed in ovulation induction, oocyte retrieval, fertilization capability and embryonic development. However, the end point which is to improve implantation and pregnancy rates after transferring embryos, remains below physiological expectations. It has been estimated that clinical implantation in the human is efficient in no more than 30% of cases considering that only one embryo is present in natural cycles, which gives us a 30% implantation rate.

A frequent pitfall found in the literature is the consideration that implantation is the result of good embryonic quality. Although this is completely true, it is not the only truth because the maternal endometrium is at least of equal relevance. In ovum donation, the endometrial factor could also be improved by individualizing the implantation window in each patient. In this proposed research we will analyze suggested markers of endometrial receptivity in order to optimize human implantation in patients undergoing assisted reproductive technologies focusing on improving endometrial receptivity in IVF and ovum donation patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for IVF or OD

Exclusion Criteria:

* Cervical stenosis

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08

PRIMARY OUTCOMES:
embryo implantation | 1 MONTH

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Revel, MD, Principal Investigator — Hadassah

REFERENCES:
- [Background] Achache H, Revel A. Endometrial receptivity markers, the journey to successful embryo implantation. Hum Reprod Update. 2006 Nov-Dec;12(6):731-46. doi: 10.1093/humupd/dml004. Epub 2006 Sep 18. PMID 16982667